CLINICAL TRIAL: NCT04982653
Title: Incisional Hernia Prevention After Open Hepatectomy by Small Tissue Bite Fascial Closure: A Randomized Clinical Trial
Brief Title: Short Stitch Versus Traditional Suture for the Prevention of Incisional Hernia After Open Hepatectomy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2021-0254; NCI-2021-04402 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2021-0254 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-06-18; First posted 2021-07-29 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Liver and Intrahepatic Bile Duct Neoplasm; Metastatic Malignant Neoplasm in the Liver; Primary Malignant Liver Neoplasm
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (hepatectomy using small bites fascial closure) (Experimental): Patients undergo hepatectomy as planned using small bites fascial method for abdominal wall closure.
  Interventions: Other: Quality-of-Life Assessment; Procedure: Surgical Procedure
- Arm II (hepatectomy using conventional fascial method) (Active Comparator): Patients undergo hepatectomy as planned using conventional fascial method for abdominal wall closure.
  Interventions: Other: Quality-of-Life Assessment; Procedure: Surgical Procedure

INTERVENTIONS:
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Procedure: Surgical Procedure — Undergo hepatectomy using small bites fascial method for abdominal wall closure
  Other Names: Operation; Surgery; Surgical; Surgical Intervention; Surgical Interventions; Surgical Procedures; Type of Surgery
  Arms: Arm I (hepatectomy using small bites fascial closure)
Procedure: Surgical Procedure — Undergo hepatectomy using conventional fascial method for abdominal wall closure
  Other Names: Operation; Surgery; Surgical; Surgical Intervention; Surgical Interventions; Surgical Procedures; Type of Surgery
  Arms: Arm II (hepatectomy using conventional fascial method)

SUMMARY:
This clinical trial compares two different kinds of surgical closing techniques, short stitch suture or traditional suture, in patients who are having liver tumor surgery. This study may help researchers learn if one technique can lower the chances of developing a hole in the wall of the abdomen (an abdominal hernia) at the incision site better than the other.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess whether small bites abdominal wall closure reduces the risk of developing incisional hernia following liver surgery.

SECONDARY OBJECTIVES:

I. To compare short-term perioperative outcomes between small bites and typical fascial closure technique.

II. To assess the hernia incidence rate of short stich versus (vs.) standard closure in subgroups of patients with inverted-L or midline incisions.

III. To assess the hernia incidence rate of Kawaguchi-Gayet hepatectomy complexity classifications I/II vs. III (hernia rate by extent of hepatectomy).

IV. To assess the hernia incidence rate of preoperative chemotherapy or no preoperative chemotherapy (hernia rate by exposure to preoperative chemotherapy).

V. To assess impact of small bites abdominal wall closure on health care quality of life following liver surgery.

VI. To assess safety of small tissue bites fascial closure suture technique versus conventional fascial closure following hepatectomy.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I (INTERVENTION): Patients undergo hepatectomy as planned using small bites fascial method for abdominal wall closure.

ARM II (CONTROL): Patients undergo hepatectomy as planned using conventional fascial method for abdominal wall closure.

After completion of study, patients are followed up at 1-4 weeks, and then at 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing hepatectomy for malignant diagnosis (primary or secondary) from 5/1/2021 through 11/1/2024 will be eligible for inclusion in this study
* Elective surgery
* Age >= 18
* Planned midline laparotomy incision or inverted-L incision

Exclusion Criteria:

* Pre-existing abdominal hernia
* History of mesh placement at prior laparotomy
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-01-04 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Radiographic incidence rate of incisional hernia | Up to 12 months after surgery
  Definition of incisional hernia will be based on the European Hernia Society: Any abdominal wall gap with or without a bulge in the area of a postoperative scar perceptible or palpable by clinical examination or imaging. Assessment of the primary outcome will occur at 3, 6, and 12 months with a computed tomography scan/magnetic resonance imaging. Scans will be read and assessed for incisional hernia by 3 independent assessors blinded to the allocation. A correlation coefficient will be determined for their assessments. The cumulative incidence rate of incisional hernia at 12 months will be estimated, along with the 95% confidence interval.

SECONDARY OUTCOMES:
Surgical site infection | Up to 90 days after surgery
Surgical site occurrence | Up to 90 days after surgery
Surgical site occurrence requiring procedural intervention | Up to 90 days after surgery
Postoperative complications | Up to 90 days after surgery
  Post-operative infection, complication or pain will be assessed using Chi-squared test or Fisher's exact test.
Need for reoperation | Up to 90 days after surgery
Need for reoperation secondary to complication of abdominal closure | Up to 90 days after surgery
Length of hospital stay (postoperatively) | Up to 90 days after surgery
  Will be compared between the two arms using two-sample t-test or Wilcoxon rank sum test.
Any readmission related to hernia repair | Up to 30 days after surgery
Health-related quality of life assessment | Up to 12 months after surgery
  Will use linear mixed effect modeling to assess the effects of time, arm as well as the interaction between arm and time.
Incidence of adverse events (AEs) | Up to 90 days after surgery
  Will be summarized using descriptive statistics (frequency, percentage) by arm, AE type, severity and attribution.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy E Newhook, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org